CLINICAL TRIAL: NCT00742040
Title: Rapid Versus Prolonged Inpatient Up-Titration of Captopril: A Randomized Clinical Trial
Brief Title: Rapid Versus Prolonged Inpatient Up-Titration of Captopril
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Paul Kantor/Principal Investigator, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1000012229
Record Dates: First submitted 2008-08-26; First posted 2008-08-27 (Estimated); Last update posted 2008-08-27 (Estimated); Status verified 2008-08

CONDITIONS: Heart Disease
Keywords: up-titration; captopril; pediatric; cardiac patients
MeSH Terms: conditions — Heart Diseases | interventions — Captopril

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Captopril
- 2 (Active Comparator)
  Interventions: Drug: Captopril

INTERVENTIONS:
Drug: Captopril — A rapid 3-day up-titration protocol
  Arms: 1
Drug: Captopril — A slower 9-day up-titration protocol
  Arms: 2

SUMMARY:
The primary objective of this study is to establish a safe and effective method of up-titration of captopril for hospital inpatients.

DETAILED DESCRIPTION:
Angiotensin converting enzyme inhibitors (ACEi) are one of the most frequently prescribed pediatric cardiac medication and overall their safety in children is widely accepted. Pediatric formulary recommendations for ACEi suggest starting with a low initial dose (0.1 mg/kg), to avoid hypotension, and up-titration for a maintenance dose. However, side ranges are quoted for maintenance doses and no guidance is given as to the best method of up-titration, The physician is left uncertain of the optimal dose and how best to achieve it.

The ultimate goal of this study is to be in a position to provide physicians caring for children with heart disease information about how to safely up-titrate this widely used medication, and by doing so to improve dosing in the wider pediatric population.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric cardiology in-patients at The Hospital for Sick Children
* Primary physician has decided to commence ACEi (the division has agreed that our institutional choice will be to start patients on captopril and up-titrate to optimal dose before converting to other ACEi)
* Patients who have been initiated on captopril within the prior 24 hours, but have not yet started up-titration, will be eligible to be randomized

Exclusion Criteria:

* Known sensitivity to ACEi
* Infants on the neonatal intensive care unit
* Treatment with any ACEi for more than 24 hours within the preceding 6 months
* Age > 18 years

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2008-08; Primary Completion 2009-08 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
The number of patients reaching a target dose of 1mg/kg/dose (given three times a day). | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Paul Kantor, MD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Roche SL, Timberlake K, Manlhiot C, Balasingam M, Wilson J, George K, McCrindle BW, Kantor PF. Angiotensin-Converting Enzyme Inhibitor Initiation and Dose Uptitration in Children With Cardiovascular Disease: A Retrospective Review of Standard Clinical Practice and a Prospective Randomized Clinical Trial. J Am Heart Assoc. 2016 May 20;5(5):e003230. doi: 10.1161/JAHA.116.003230. PMID 27207965